CLINICAL TRIAL: NCT04197973
Title: Association Between Self-reported Web-based Simple Clinical Colitis Activity Index(SCCAI) and Health-related Quality of Life Index in Patients With Ulcerative Colitis
Brief Title: Association Between Self-reported Web-based SCCAI and Health-related Quality of Life Index in UC Patients
Acronym: UC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: YooJin Lee (Other)
Collaborators: Inje University (Other); Gangnam Severance Hospital (Other); Jeju National University Hospital (Other); Soonchunhyang University Hospital (Other)
Responsible Party: Sponsor-Investigator, YooJin Lee, Professor, Keimyung University Dongsan Medical Center
Organization: Keimyung University Dongsan Medical Center (Other)
Other Study IDs: 2018-05-056
Record Dates: First submitted 2019-11-29; First posted 2019-12-13 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Quality of Life; Ulcerative Colitis
Keywords: SCCAI; health-related quality of life index
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An accurate assessment of disease activity is crucial for the treatment of patients with ulcerative colitis (UC). Recent studies have reported that the Simple Clinical Colitis Activity Index (SCCAI) correlates well with Mayo score. A recent report demonstrated that SCCAI has a significant correlation with the degree of health-related quality of life in UC patients. It is also reported that the self-administered SCCAI through the web-based input tool at home is highly correlated with the SCCAI assessed by physician. The aim of this study was to investigate the relationship between self-administered web-based SCCAI and the health-related quality of life of UC patients.

DETAILED DESCRIPTION:
An accurate assessment of disease activity is crucial for the treatment of patients with ulcerative colitis (UC). Several indices have been used to assess disease activity in patients with UC. Mayo score is the most widely used index for UC activity measurement. Meanwhile, recent studies have reported that the Simple Clinical Colitis Activity Index (SCCAI) correlates well with Mayo score. SCCAI is consisted of only clinical items and includes items such as nocturnal diarrhea and urgent defecation which are more closely related to the quality of life of patients. In this regard, a recent report demonstrated that SCCAI has a significant correlation with the degree of health-related quality of life in UC patients.

Since SCCAI is composed of only clinical parameters, it can be evaluated by the patients themselves. According to recent research, the self-administered SCCAI was reported to have a high correlation with the SCCAI assessed by physician (correlation coefficient = 0.79). Moreover, it is also reported that the self-administered SCCAI through the web-based input tool at home is highly correlated with the SCCAI assessed by physician (Spearman's correlation = 0.79). These results suggest that the patient's self-reported SCCAI can be applied to actual clinical practice, and it will enable remote monitoring and flexible follow-up depending on the patient's disease activity. If self-administered SCCAI is to be applied as a more valid disease activity assessment tools, it also properly reflects patient's quality of life status. However, it is not yet known whether the self-administered SCCAI using web-based tools reflects the quality of life of patients.

The aim of this study was to investigate the relationship between self-administered web-based SCCAI and the health-related quality of life of UC patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of UC for >3 months
* familiarity with online communication (e.g., use of the Internet)
* Consent for study participation

Exclusion Criteria:

* Previous colon resection or other UC related bowel surgery
* Psychiatric or intellectual disability
* Lack of ability for access or use online tools

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with ulcerative colitis visiting Inje University College of Medicine Ilsan Paik Hospital, Gangnam Severance Hospital, Jeju National University Hospital, Keimyung University Dongsan Medical Center, Soonchunhyang University Hospital Cheonan will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2019-12-18 (Actual); Primary Completion 2020-12-20 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between SCCAI and health-related quality of life (IBD-Q 32) in patient with UC | Baseline
  Correlation between SCCAI administered by a web-based input tool at home and health-related quality of life (IBD-Q 32) in patient with UC
Correlation between SCCAI and health-related quality of life (IBD-Q 32) in patient with UC | 3 months after baseline
  Correlation between SCCAI administered by a web-based input tool at home and health-related quality of life (IBD-Q 32) in patient with UC
Correlation between SCCAI and health-related quality of life (IBD-Q 32) in patient with UC | 6 months after baseline
  Correlation between SCCAI administered by a web-based input tool at home and health-related quality of life (IBD-Q 32) in patient with UC

SECONDARY OUTCOMES:
Correlation between self-administered SCCAI and SCCAI assessed by physician | Baseline
  Correlation between SCCAI administered by a web-based input tool at home and SCCAI assessed by physician
Correlation between self-administered SCCAI and SCCAI assessed by physician | 3 months after baseline
  Correlation between SCCAI administered by a web-based input tool at home and SCCAI assessed by physician
Correlation between self-administered SCCAI and SCCAI assessed by physician | 6 months after baseline
  Correlation between SCCAI administered by a web-based input tool at home and SCCAI assessed by physician

CONTACTS AND LOCATIONS:
Overall Officials: Yoo Jin Lee, Professor, Study Director — Keimyung University Dongsan Medical Center
Locations (1):
- KeimyungUniversity, Daegu, Dalseo-gu, South Korea